CLINICAL TRIAL: NCT03799627
Title: Phase 2, Randomized, Open-Label, Active-Controlled, Efficacy, Safety, Pharmacokinetics, and Pharmacodynamics Study of Oral Vadadustat for the Treatment of Anemia in Hemodialysis Subjects Converting From Epoetin Alfa (FO2RWARD-2)
Brief Title: Study of Vadadustat in Hemodialysis Participants With Anemia Switching From Epoetin Alfa
Acronym: FO2RWARD-2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Akebia Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AKB-6548-CI-0025
Record Dates: First submitted 2018-12-03; First posted 2019-01-10 (Actual); Results first posted 2022-09-29 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: Anemia; Dialysis-dependent Chronic Kidney Disease
Keywords: Vadadustat; AKB-6548; Anemia; Chronic kidney disease (CKD); erythropoietin
MeSH Terms: conditions — Anemia; Renal Insufficiency, Chronic | interventions — vadadustat; Epoetin Alfa

STUDY DESIGN:
Intervention Model Description: Randomized, Open-Label, Active-Controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Vadadustat (Experimental): The initial dose of Vadadustat (300, 450, or 600 milligrams [mg]) will be based upon the dose of Epoetin Alfa dose participants had received prior to Vadadustat treatment
  Interventions: Drug: Vadadustat
- Vadadustat TIW (Experimental): Participants randomized to Vadadustat (Main and erythropoiesis-stimulating agent [ESA] hyporesponder parallel studies) who complete a once-daily dosing regimen treatment period and meet eligibility criteria for transition to three times weekly (TIW) dosing will switch to TIW dosing
  Interventions: Drug: Vadadustat TIW
- Epoetin Alfa (Active Comparator): Epoetin Alfa
  Interventions: Drug: Epoetin Alfa

INTERVENTIONS:
Drug: Vadadustat — Vadadustat Tablets 150 mg
  Other Names: AKB-6548
  Arms: Vadadustat
Drug: Epoetin Alfa — Epoetin Alfa
  Other Names: Procrit; Epogen
  Arms: Epoetin Alfa
Drug: Vadadustat TIW — Oral Vadadustat
  Arms: Vadadustat TIW

SUMMARY:
This is a Phase 2 open-label efficacy, safety, and pharmacokinetic/pharmacodynamic (PK/PD) study to evaluate oral Vadadustat for the treatment of anemia in hemodialysis participants converting from Epoetin Alfa therapy.

DETAILED DESCRIPTION:
This is a Phase 2, randomized, open-label study to evaluate efficacy and safety of oral Vadadustat for the treatment of anemia in hemodialysis participants converting from Epoetin Alfa therapy. The study will be conducted in two parts running in parallel: Part 1, Main Study in a hemodialysis population on maintenance treatment with Epoetin Alfa; Part 2 is in a hemodialysis population that are erythropoiesis-stimulating agent (ESA) hyporesponders on maintenance treatment with Epoetin Alfa. For all participants (Main and ESA hyporesponder parallel study), the study will include a Screening Period, a Treatment Period, and a Safety Follow-Up Period. PK and PD sampling will be done throughout the study. The aim is to achieve and maintain hemoglobin (Hb) levels within the target range of 10.0 to 11.0 grams per deciliter (g/dL), inclusive, while targeting the middle of the range and minimizing excursions outside the target range.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age, providing informed consent
* Receiving chronic, outpatient in-center hemodialysis (TIW) for end-stage renal disease for at least 12 weeks prior to Screening
* Maintained on intravenous Epoetin Alfa therapy for 8 weeks prior to and including Screening through Screening Visit 2 (SV2)
* Eligibility in the Main study and erythropoiesis-stimulating agent (ESA) hyporesponder parallel study is based on the following mean weekly Epoetin Alfa doses:

  1. Main study: Mean weekly Epoetin Alfa dose <300 Units per kilogram per week (U/kg/week) for 8 weeks prior to SV2;
  2. ESA hyporesponder parallel study: Mean weekly Epoetin Alfa dose ≥300 U/kg/week for 8 weeks prior to SV2
* Two Hb values measured by the central laboratory at least 4 days apart between Screening Visit 1 (SV1) and SV2 as indicated:.

  1. Main study: 2 Hb values between 8.5 and 11.0 g/dL, inclusive;
  2. ESA hyporesponder parallel study: 2 Hb values between 8.0 and 10.0 grams per deciliter (g/dL), inclusive
* Serum ferritin ≥100 nanograms per milliliter (ng/mL) and transferrin saturation (TSAT) ≥20% during Screening
* Folate and vitamin B12 measurements ≥ lower limit of normal during Screening
* Hemodialysis adequacy as indicated by single-pool Kt/Vurea ≥1.2 using the most recent historical measurement within 8 weeks prior to or during Screening
* Understands the procedures and requirements of the study and provides written informed consent and authorization for protected health information disclosure

Exclusion Criteria:

* Anemia due to a cause other than chronic kidney disease (e.g., sickle cell disease, myelodysplastic syndromes, bone marrow fibrosis, hematologic malignancy, myeloma, hemolytic anemia, thalassemia, or pure red cell aplasia)
* Active bleeding or recent blood loss within 8 weeks prior to randomization
* Red blood cell (RBC) transfusion within 8 weeks prior to randomization
* Anticipated to discontinue hemodialysis during the study
* Judged by the Investigator that the participant is likely to need rescue therapy (ESA administration or RBC transfusion) immediately after enrollment in the study
* History of chronic liver disease (e.g., chronic infectious hepatitis, chronic autoimmune liver disease, cirrhosis or fibrosis of the liver)
* Aspartate aminotransferase (AST)/serum glutamic oxaloacetic transaminase (SGOT), alanine aminotransferase (ALT)/serum glutamic pyruvic transaminase (SGPT), or total bilirubin >1.5 x upper limit of normal (ULN) during Screening. Participants with a history of Gilbert's syndrome are not excluded.
* Current uncontrolled hypertension as determined by the Investigator that would contraindicate the use of Epoetin Alfa
* Acute coronary syndrome (hospitalization for unstable angina or myocardial infarction), surgical or percutaneous intervention for coronary, cerebrovascular or peripheral artery disease (aortic or lower extremity), surgical or percutaneous valvular replacement or repair, sustained ventricular tachycardia, hospitalization for heart failure (HF) or New York Heart Association Class IV HF, or stroke within 12 weeks prior to or during Screening
* History of new or recurrent malignancy within 2 years prior to and during Screening or currently receiving treatment or suppressive therapy for cancer. Participants with treated basal cell carcinoma of skin, curatively resected squamous cell carcinoma of skin, or cervical carcinoma in situ are not excluded.
* History of deep vein thrombosis or pulmonary embolism within 12 weeks prior to or during Screening
* History of hemosiderosis or hemochromatosis
* History of prior organ transplantation (participants with a history of failed kidney transplant or corneal transplants are not excluded)
* Scheduled organ transplant from a living donor and participants on the kidney transplant wait-list who are expected to receive a transplant within 6 months
* History of a prior hematopoietic stem cell or bone marrow transplant (stem cell therapy for knee arthritis is not excluded)
* Known hypersensitivity to Vadadustat, Epoetin Alfa, or any of their excipients
* Any prior use of a hypoxia-inducible factor prolyl-hydroxylase (HIF-PH) inhibitor or any use of an investigational medication within 30 days or 5 half-lives of the investigational medication (whichever is longer), prior to randomization
* For female participants of non-childbearing potential:

  1. inability to confirm surgical sterility (e.g., hysterectomy, bilateral tubal ligation, bilateral oophorectomy) at least 1 month prior to Screening;
  2. not considered post-menopausal (no menses for >1 year with follicle stimulating hormone >40 U/Liter at Screening)
* For female participants of childbearing potential:

  1. lack of confirmation of the use of acceptable forms of contraception* for a minimum of one complete menstrual cycle prior to Screening;
  2. positive serum pregnancy test at SV2;
  3. unwilling to use two acceptable forms of contraception* (at least one of which must be a barrier method) starting Baseline/Day 1, throughout the Treatment Period and for 30 days after the final study drug administration
* Breastfeeding during Screening or throughout the Treatment Period and for 30 days after the final study drug administration
* Donation of ova starting at Screening, throughout the Treatment Period, and for 30 days after the final study drug administration
* Male participants who have not had a vasectomy and do not agree to the following: use of an acceptable form of contraception* during the study and for 30 days after the last dose of the study drug; to not donate semen during the study and for at least 30 days after the last dose of Vadadustat
* Participants with bilateral native nephrectomy
* Any other reason, which in the opinion of the Investigator, would make the participant not suitable for participation in the study

  * Acceptable forms of contraception include:

    * Established use of oral, injected or implanted hormonal methods of contraception;
    * Placement of an intrauterine device or intrauterine system;
    * Barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2019-01-31 (Actual); Primary Completion 2020-06-05 (Actual); Study Completion 2020-07-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Director — Akebia Therapeutics Inc.
Locations (37):
- United States (37):
  - Research Site, Fresno, California
  - Research Site, Granada Hills, California
  - Research Site, Los Angeles, California
  - Research Site, Northridge, California
  - Research Site, Riverside, California
  - Research Site #1, San Dimas, California
  - Research Site #2, San Dimas, California
  - Research Site, San Gabriel, California
  - Research Site, Tarzana, California
  - Research Site, Vacaville, California
  - Research Site, Victorville, California
  - Research Site, Denver, Colorado
  - Research Site, Bridgeport, Connecticut
  - Research Site, Hartford, Connecticut
  - Research Site, Coral Gables, Florida
  - Research Site, Hollywood, Florida
  - Research Site, Miami, Florida
  - Research Site, Tampa, Florida
  - Research Site, Winter Park, Florida
  - Research Site, Augusta, Georgia
  - Research Site, Statesboro, Georgia
  - Research Site, Roseville, Michigan
  - Research Site #1, Minneapolis, Minnesota
  - Research Site #2, Minneapolis, Minnesota
  - Research Site, Kansas City, Missouri
  - Research Site, Las Vegas, Nevada
  - Research Site, The Bronx, New York
  - Research Site, Asheville, North Carolina
  - Research Site, Wilmington, North Carolina
  - Research Site, Canton, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, El Paso, Texas
  - Research Site, Houston, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Chesapeake, Virginia
  - Research Site, Norfolk, Virginia
  - Research Site, Wauwatosa, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Natale P, Palmer SC, Jaure A, Hodson EM, Ruospo M, Cooper TE, Hahn D, Saglimbene VM, Craig JC, Strippoli GF. Hypoxia-inducible factor stabilisers for the anaemia of chronic kidney disease. Cochrane Database Syst Rev. 2022 Aug 25;8(8):CD013751. doi: 10.1002/14651858.CD013751.pub2. PMID 36005278

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 540 participants were screened, of which 175 participants were enrolled and randomized into the 2 parts of this study (Main Study; n=165; Erythropoiesis-stimulating Agent (ESA) Hyporesponder Parallel Study: n=10). A total of 365 participants failed screening. Participants were randomized to either a Vadadustat or Epoetin Alfa treatment group, and randomization was stratified by mean weekly Epoetin Alfa dose calculated over a period of 8 weeks prior to Screening Visit 2.
Groups:
- Low Dose of Epoetin Alfa: Vadadustat 300 mg: Participants who were maintained on the low dose of Epoetin Alfa (≤90 units per kilogram per week [U/kg/week]) prior to and including the Screening Period for a minimum of 8 weeks prior to Screening Visit 2 were administered an oral dose of Vadadustat 300 milligram (mg) tablet per day (QD) until Week 12. Eligible participants based on investigator's discretion were switched from daily dosing to three times per week (TIW) dosing of the starting Vadadustat dose (300 mg) plus a 150 mg greater dose (450 mg) to maintain target hemoglobin (Hb) levels during Week 12 to Week 14. Non-eligile participants continued with daily dosing. Participants who reported a decline in Hb ≥0.5 grams per deciliter (g/dL) were eligible for a dose increase by another 150 mg until Week 20.
- Low Dose of Epoetin Alfa: Vadadustat 450 mg: Participants who were maintained on the low dose of Epoetin Alfa (≤90 U/kg/week) prior to and including the Screening Period for a minimum of 8 weeks prior to Screening Visit 2 were administered an oral dose of Vadadustat 450 mg tablet QD until Week 12. Eligible participants based on investigator's discretion were switched from daily dosing to TIW dosing of the starting Vadadustat dose (450 mg) plus a 150 mg greater dose (600 mg) to maintain target Hb levels during Week 12 to Week 14. Non-eligible participants continued with daily dosing. Participants who reported a decline in Hb ≥0.5 g/dL were eligible for a dose increase by another 150 mg until Week 20.
- Low Dose of Epoetin Alfa: Epoetin Alfa: Participants who were maintained on the low dose of Epoetin Alfa (≤90 U/kg/week) prior to and including the Screening Period were administered TIW dosing of Epoetin Alfa for the entire Treatment Period based on the participant's Hb value and the approved Epoetin Alfa United States (US) Package Insert (PI) for adult participants with chronic kidney disease (CKD) on dialysis. The dose was adjusted to achieve and maintain target Hb levels of 10.0-11.0 g/dL, inclusive.
- High Dose of Epoetin Alfa: Vadadustat 300 mg: Participants who were maintained on the high dose of Epoetin Alfa (>90 to <300 U/kg/week) prior to and including the Screening Period for a minimum of 8 weeks prior to Screening Visit 2 were administered an oral dose of Vadadustat 300 mg tablet QD until Week 12. Eligible participants based on investigator's discretion were switched from daily dosing to TIW dosing of the starting Vadadustat dose (300 mg) plus a 150 mg greater dose (450 mg) to maintain target Hb levels during Week 12 to Week 14. Non-eligible participants continued with daily dosing. Participants who reported a decline in Hb ≥0.5 g/dL were eligible for a dose increase by another 150 mg until Week 20.
- High Dose of Epoetin Alfa: Vadadustat 450 mg: Participants who were maintained on the high dose of Epoetin Alfa (>90 to <300 U/kg/week) prior to and including the Screening Period for a minimum of 8 weeks prior to Screening Visit 2 were administered an oral dose of Vadadustat 450 mg tablet QD until Week 12. Eligible participants based on investigator's discretion were switched from daily dosing to TIW dosing of the starting Vadadustat dose (450 mg) plus a 150 mg greater dose (600 mg) to maintain target Hb levels during Week 12 to Week 14. Non-eligible participants continued with daily dosing. Participants who reported a decline in Hb ≥0.5 g/dL were eligible for a dose increase by another 150 mg until Week 20.
- High Dose of Epoetin Alfa: Vadadustat 600 mg: Participants who were maintained on the high dose of Epoetin Alfa (>90 to <300 U/kg/week) prior to and including the Screening Period for a minimum of 8 weeks prior to Screening Visit 2 were administered an oral dose of Vadadustat 600 mg tablet QD until Week 12. Eligible participants based on investigator's discretion were switched from daily dosing to TIW dosing of the starting Vadadustat dose (600 mg) plus a 150 mg greater dose (750 mg) to maintain target Hb levels during Week 12 to Week 14. Non-eligible participants continued with daily dosing. Participants who reported a decline in Hb ≥0.5 g/dL were eligible for a dose increase by another 150 mg until Week 20.
- High Dose of Epoetin Alfa: Epoetin Alfa: Participants who were maintained on the high dose of Epoetin Alfa (>90 to <300 U/kg/week) prior to and including the Screening Period were administered TIW dosing of Epoetin Alfa for the entire Treatment Period based on the participant's Hb value and the approved Epoetin Alfa US PI for adult participants with CKD on dialysis. The dose was adjusted to achieve and maintain target Hb levels of 10.0-11.0 g/dL, inclusive.
- ESA Hyporesponder: Vadadustat 600 mg: In the Erythropoiesis-stimulating Agent (ESA) Hyporesponder Parallel Study, participants who were maintained on a ≥300 U/kg/week dose of Epoetin Alfa prior to and including the Screening Period for a minimum of 8 weeks prior to Screening Visit 2 were administered an oral dose of Vadadustat 600 mg tablet QD until Week 12. Eligible participants based on investigator's discretion were switched from daily dosing to TIW dosing of the starting Vadadustat dose (600 mg) plus a 150 mg greater dose (750 ng) to maintain target Hb levels during Week 12 to Week 14. Non-eligible participants continued with daily dosing. Participants who reported a decline in Hb ≥0.5 g/dL were eligible for a dose increase by another 150 mg until Week 20.
- ESA Hyporesponder: Epoetin Alfa: In the ESA Hyporesponder Parallel Study, participants who were maintained on a ≥300 U/kg/week dose of Epoetin Alfa prior to and including the Screening Period for a minimum of 8 weeks prior to Screening Visit 2 were administered TIW dosing of Epoetin Alfa based on the participant's central laboratory Hb value and the approved Epoetin Alfa US PI for adult participants with CKD on dialysis. The dose was adjusted to achieve and maintain target Hb levels of 10.0-11.0 g/dL, inclusive.
Period: Overall Study
Arm/Group | Low Dose of Epoetin Alfa: Vadadustat 300 mg | Low Dose of Epoetin Alfa: Vadadustat 450 mg | Low Dose of Epoetin Alfa: Epoetin Alfa | High Dose of Epoetin Alfa: Vadadustat 300 mg | High Dose of Epoetin Alfa: Vadadustat 450 mg | High Dose of Epoetin Alfa: Vadadustat 600 mg | High Dose of Epoetin Alfa: Epoetin Alfa | ESA Hyporesponder: Vadadustat 600 mg | ESA Hyporesponder: Epoetin Alfa
Started | 35 | 34 | 23 | 18 | 21 | 21 | 13 | 5 | 5
Completed | 27 | 23 | 22 | 8 | 12 | 8 | 10 | 3 | 2
Not Completed | 8 | 11 | 1 | 10 | 9 | 13 | 3 | 2 | 3
Not completed — Adverse Event | 1 | 2 | 0 | 0 | 2 | 5 | 0 | 2 | 0
Not completed — Physician Decision | 2 | 2 | 0 | 0 | 2 | 2 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 2 | 0 | 3 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Not completed — Death | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Study Drug Put on Hold | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Due to Urgent Safety Measures Letter | 1 | 2 | 0 | 2 | 1 | 0 | 0 | 0 | 0
Not completed — Kidney Transplantation | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Participant Was on Rescue Epogen | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Not completed — Placed on Dose Hold Until End of Treatment | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Met Exclusion Criteria | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Investigational Product Noncompliance | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Participant Relocation | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Not completed — Eurofin Issue | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Noncompliance with Site Instructions | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Participant's Last Dose Prior to End of Treatment | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Changes In Hemoglobin Values | 1 | 2 | 1 | 0 | 0 | 2 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Dose of Epoetin Alfa: Vadadustat 300 mg | Low Dose of Epoetin Alfa: Vadadustat 450 mg | Low Dose of Epoetin Alfa: Epoetin Alfa | High Dose of Epoetin Alfa: Vadadustat 300 mg | High Dose of Epoetin Alfa: Vadadustat 450 mg | High Dose of Epoetin Alfa: Vadadustat 600 mg | High Dose of Epoetin Alfa: Epoetin Alfa | ESA Hyporesponder: Vadadustat 600 mg | ESA Hyporesponder: Epoetin Alfa | Total
Number analyzed (Participants) | 35 | 34 | 23 | 18 | 21 | 21 | 13 | 5 | 5 | 175
Age, Customized [Count of Participants; unit: Participants]
  <65 years | 20 | 22 | 15 | 11 | 18 | 13 | 7 | 4 | 3 | 113
  >=65 years | 15 | 12 | 8 | 7 | 3 | 8 | 6 | 1 | 2 | 62
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 13 | 4 | 7 | 7 | 9 | 6 | 4 | 3 | 67
  Male | 21 | 21 | 19 | 11 | 14 | 12 | 7 | 1 | 2 | 108
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 4
  Asian | 2 | 1 | 1 | 1 | 1 | 1 | 1 | 0 | 1 | 9
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 4
  Black or African American | 18 | 19 | 7 | 8 | 13 | 14 | 6 | 2 | 2 | 89
  White | 10 | 9 | 13 | 5 | 6 | 5 | 5 | 3 | 0 | 56
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 4 | 4 | 1 | 2 | 1 | 0 | 1 | 0 | 0 | 13

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Hemoglobin (Hb) Between Baseline and the Primary Evaluation Period (PEP)
Description: Change from Baseline in Hb value was calculated as the PEP Hb value minus the Baseline Hb value. The PEP value was the average Hb value from Week 10 to Week 12. The Baseline Hb value was defined as the average of the final two Hb values prior to start of dosing on Day 1.
Time Frame: Baseline; Week 10 to Week 12
Population: Randomized Population: All randomized participants. Analysis of this population was based on the randomized treatment.
Measure: Mean (Standard Deviation); unit: grams per deciliter (g/dL)
Arm/Group | Low Dose of Epoetin Alfa: Vadadustat 300 mg | Low Dose of Epoetin Alfa: Vadadustat 450 mg | Low Dose of Epoetin Alfa: Epoetin Alfa | High Dose of Epoetin Alfa: Vadadustat 300 mg | High Dose of Epoetin Alfa: Vadadustat 450 mg | High Dose of Epoetin Alfa: Vadadustat 600 mg | High Dose of Epoetin Alfa: Epoetin Alfa | ESA Hyporesponder: Vadadustat 600 mg | ESA Hyporesponder: Epoetin Alfa
Number analyzed (Participants) | 35 | 34 | 23 | 18 | 21 | 21 | 13 | 5 | 5
grams per deciliter (g/dL)
  Baseline | 10.223 (0.5805) | 10.059 (0.6769) | 10.165 (0.6806) | 9.778 (0.6832) | 10.288 (0.5445) | 10.095 (0.7150) | 9.950 (0.7950) | 9.530 (0.2864) | 9.620 (0.6925)
  Change from Baseline at PEP: number analyzed (Participants) | 30 | 30 | 23 | 12 | 18 | 14 | 12 | 4 | 5
  Change from Baseline at PEP | -0.371 (0.8920) | 0.072 (1.1353) | 0.160 (0.7519) | -0.911 (1.3515) | -0.284 (1.0383) | -0.418 (1.2752) | 0.268 (1.0087) | -0.671 (0.7643) | -0.290 (1.7730)

2. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was defined as any untoward medical occurrence (including a clinically significant abnormal laboratory finding) that occurred in the protocol-specified AE reporting period. An AE included medical conditions, signs, and symptoms not previously observed in the participant that emerged during the protocol-specified AE reporting period, including signs or symptoms associated with pre-existing underlying conditions that were not present prior to the AE reporting period. TEAEs, defined as AEs that began (or pre-existing AEs that worsened) on or after the first dose through each participant's last participation date, are reported.
Time Frame: Up to Week 24
Population: Safety Population: all participants in the Randomized Population who received at least 1 dose of study drug. Analysis of this population was based on actual treatment received. Participants who received Vadadustat and Epoetin Alfa in error were classified by the more frequently received drug. One participant randomized to the Low Dose of Epoetin Alfa: Vadadustat 300 mg arm inadvertently received 450 mg of Vadadustat.
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose of Epoetin Alfa: Vadadustat 300 mg | Low Dose of Epoetin Alfa: Vadadustat 450 mg | Low Dose of Epoetin Alfa: Epoetin Alfa | High Dose of Epoetin Alfa: Vadadustat 300 mg | High Dose of Epoetin Alfa: Vadadustat 450 mg | High Dose of Epoetin Alfa: Vadadustat 600 mg | High Dose of Epoetin Alfa: Epoetin Alfa | ESA Hyporesponder: Vadadustat 600 mg | ESA Hyporesponder: Epoetin Alfa
Number analyzed (Participants) | 34 | 35 | 23 | 18 | 21 | 21 | 13 | 5 | 5
Participants | 18 | 27 | 13 | 12 | 14 | 13 | 9 | 5 | 3

3. Primary Outcome: Number of Participants With Clinically Significant Changes From Baseline in Laboratory Parameter Values
Description: Parameters assessed for laboratory values included hematology (excluding the primary and secondary efficacy endpoint results related to Hb), clinical chemistry, lipid profiles, and glucose. The investigator was responsible for reviewing laboratory results for clinically significant changes.
Time Frame: Up to Week 24
Population: Safety Population. Analysis of this population was based on the actual treatment received. Participants who received Vadadustat and Epoetin Alfa in error were classified by the more frequently received drug. One participant randomized to the Low Dose of Epoetin Alfa: Vadadustat 300 mg arm inadvertently received 450 mg of Vadadustat.
Measure: Count of Participants; unit: Participants
Groups:
- Low Dose of Epoetin Alfa: Epoetin Alfa: Participants who were maintained on the low dose of Epoetin Alfa (≤90 U/kg/week) prior to and including the screening period for a minimum of 8 weeks prior to screening visit 2, were administered with three times a week (TIW) dose of Epoetin Alfa based on the participant's central laboratory hemoglobin (Hb) value and the approved Epoetin Alfa United States (US) Package Insert (PI) for adult participants with CKD on dialysis. Dose was adjusted to achieve and maintain Hb levels within the target range of 10.0 and 11.0 g/dL, inclusive.
Arm/Group | Low Dose of Epoetin Alfa: Vadadustat 300 mg | Low Dose of Epoetin Alfa: Vadadustat 450 mg | Low Dose of Epoetin Alfa: Epoetin Alfa | High Dose of Epoetin Alfa: Vadadustat 300 mg | High Dose of Epoetin Alfa: Vadadustat 450 mg | High Dose of Epoetin Alfa: Vadadustat 600 mg | High Dose of Epoetin Alfa: Epoetin Alfa | ESA Hyporesponder: Vadadustat 600 mg | ESA Hyporesponder: Epoetin Alfa
Number analyzed (Participants) | 34 | 35 | 23 | 18 | 21 | 21 | 13 | 5 | 5
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Clinically Significant Changes From Baseline in Vital Sign Values
Description: Parameters assessed for vital signs included sitting (at rest for a minimum of 5 minutes) heart rate, respiratory rate, body temperature, and blood pressure. The investigator was responsible for reviewing vital sign values for clinically significant changes.
Time Frame: Up to Week 24
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose of Epoetin Alfa: Vadadustat 300 mg | Low Dose of Epoetin Alfa: Vadadustat 450 mg | Low Dose of Epoetin Alfa: Epoetin Alfa | High Dose of Epoetin Alfa: Vadadustat 300 mg | High Dose of Epoetin Alfa: Vadadustat 450 mg | High Dose of Epoetin Alfa: Vadadustat 600 mg | High Dose of Epoetin Alfa: Epoetin Alfa | ESA Hyporesponder: Vadadustat 600 mg | ESA Hyporesponder: Epoetin Alfa
Number analyzed (Participants) | 34 | 35 | 23 | 18 | 21 | 21 | 13 | 5 | 5
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Number of Participants Classified as Hb Outliers
Description: The target range for Hb was from 10.0 to 11.0 grams per deciliter (g/dL). Hb outliers included participants with a Hb increase of more than 12.0 g/dL or <8.0 g/dL and decline in Hb ≥0.5 g/dL from Baseline, and a Hb increase to more than 1.0 g/dL within any 2-week interval during the Study Period.
Time Frame: Weeks 13 - 20
Population: Safety Population. Analysis of this population was based on the actual treatment received. Participants who received Vadadustat and Epoetin Alfa in error were classified by the more frequently received drug. Only participants with available data were included in the analysis. The rows presenting data for HB > 12.0 g/dL, HB > 13.0 g/dL and HB > 14.0 g/dL are mutually exclusive.
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose of Epoetin Alfa: Vadadustat 300 mg | Low Dose of Epoetin Alfa: Vadadustat 450 mg | Low Dose of Epoetin Alfa: Epoetin Alfa | High Dose of Epoetin Alfa: Vadadustat 300 mg | High Dose of Epoetin Alfa: Vadadustat 450 mg | High Dose of Epoetin Alfa: Vadadustat 600 mg | High Dose of Epoetin Alfa: Epoetin Alfa | ESA Hyporesponder: Vadadustat 600 mg | ESA Hyporesponder: Epoetin Alfa
Number analyzed (Participants) | 30 | 27 | 23 | 10 | 16 | 13 | 12 | 3 | 5
Participants
  Hb >12.0 g/dL | 2 | 2 | 3 | 0 | 1 | 0 | 1 | 0 | 0
  Hb >13.0 g/dL | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Hb >14.0 g/dL | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Hb <8.0 g/dL and decline in Hb ≥0.5 g/dL from Baseline | 2 | 2 | 0 | 1 | 1 | 3 | 1 | 1 | 1
  Hb increase >1.0 g/dL within any 2-week interval | 4 | 8 | 4 | 4 | 2 | 3 | 6 | 0 | 2

6. Secondary Outcome: Number of Participants With Hb Values Within the Target Range at the PEP
Description: The target range for Hb was from 10.0 to 11.0 g/dL, inclusive. The PEP was comprised of Week 10 to Week 12.
Time Frame: Week 10 to Week 12
Population: Randomized Population. Analysis of this population was based on the randomized treatment. Participants with non-missing values were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose of Epoetin Alfa: Vadadustat 300 mg | Low Dose of Epoetin Alfa: Vadadustat 450 mg | Low Dose of Epoetin Alfa: Epoetin Alfa | High Dose of Epoetin Alfa: Vadadustat 300 mg | High Dose of Epoetin Alfa: Vadadustat 450 mg | High Dose of Epoetin Alfa: Vadadustat 600 mg | High Dose of Epoetin Alfa: Epoetin Alfa | ESA Hyporesponder: Vadadustat 600 mg | ESA Hyporesponder: Epoetin Alfa
Number analyzed (Participants) | 30 | 30 | 23 | 12 | 18 | 14 | 12 | 4 | 5
Participants | 12 | 13 | 15 | 1 | 4 | 4 | 6 | 0 | 0

7. Secondary Outcome: Mean Change in Hb From the PEP to the Secondary Evaluation Period (SEP) in Participants Who Transitioned to Three Times Per Week (TIW) Vadadustat Dosing After Week 12
Description: Change from PEP was calculated as the SEP value minus the PEP value. The PEP value was the average Hb value from Week 10 to Week 12. The SEP value was the average Hb value from Week 18 to Week 20. For the Main Study, analysis is presented per dose level according to the starting dose in TIW regimen, as well as being presented as a combined arm for "Vadadustat Total (TIW dosing regimen)". For the ESA Hyporesponder Parallel Study, a starting dose classification for TIW dosing regimen was not applicable due to no participants switching from Vadadustat QD to TIW dosing.
Time Frame: Week 10 to Week 12; Week 18 to Week 20
Population: Randomized Population. Analysis of this population was based on the randomized treatment. Only those who switched from Vadadustat QD to TIW dosing after Week 12 were included in the analysis (17 participants overall in Main Study and 0 participants in ESA Hyporesponder Parallel Study).
Measure: Mean (Standard Deviation); unit: g/dL
Groups:
- Vadadustat 300 mg (Starting Dose in TIW Dosing Regimen): After completing the 12-week QD dosing regimen, eligible participants based on investigator's discretion were switched from daily dosing to TIW dosing to receive a starting dose of Vadadustat 300 mg (1 tablet greater [150 mg] than final dose in QD dosing regimen [150 mg]). Participants who reported a decline in Hb ≥0.5 g/dL were eligible for a dose increase by another 150 mg until Week 20.
- Vadadustat 450 mg (Starting Dose in TIW Dosing Regimen): After completing the 12-week QD dosing regimen, eligible participants based on investigator's discretion were switched from daily dosing to TIW dosing to receive a starting dose of Vadadustat 450 mg (1 tablet greater [150 mg] than final dose in QD dosing regimen [300 mg]). Participants who reported a decline in Hb ≥0.5 g/dL were eligible for a dose increase by another 150 mg until Week 20.
- Vadadustat 600 mg (Starting Dose in TIW Dosing Regimen): After completing the 12-week QD dosing regimen, eligible participants based on investigator's discretion were switched from daily dosing to TIW dosing to receive a starting dose of Vadadustat 600 mg (1 tablet greater [150 mg] than final dose in QD dosing regimen [450 mg]). Participants who reported a decline in Hb ≥0.5 g/dL were eligible for a dose increase by another 150 mg until Week 20.
- Vadadustat 750 mg (Starting Dose in TIW Dosing Regimen): After completing the 12-week QD dosing regimen, eligible participants based on investigator's discretion were switched from daily dosing to TIW dosing to receive a starting dose of Vadadustat 750 mg (1 tablet greater [150 mg] than final dose in QD dosing regimen [600 mg]). Participants who reported a decline in Hb ≥0.5 g/dL were eligible for a dose increase by another 150 mg until Week 20.
- Vadadustat Total (TIW Dosing Regimen): After completing the 12-week QD dosing regimen, eligible participants based on investigator's discretion were switched from daily dosing to TIW dosing to receive a starting dose of Vadadustat 1 tablet greater (150 mg) than final dose in QD dosing regimen. Vadadustat Total comprises all participants who switched from Vadadustat QD to TIW dosing regimen in the Main Study (i.e., combined arm for starting doses of 300mg, 450 mg, 600 mg and 750 mg). Participants who reported a decline in Hb ≥0.5 g/dL were eligible for a dose increase by another 150 mg until Week 20.
- ESA Hyporesponder Parallel Study: Vadadustat ≤ 750 mg (TIW Dosing Regimen): After completing the 12-week QD dosing regimen, eligible participants based on investigator's discretion were switched from daily dosing to TIW dosing to receive a starting dose of Vadadustat ≤ 750 mg (1 tablet greater [150 mg] than final dose in QD dosing regimen). Participants who reported a decline in Hb ≥0.5 g/dL were eligible for a dose increase by another 150 mg until Week 20.
Arm/Group | Vadadustat 300 mg (Starting Dose in TIW Dosing Regimen) | Vadadustat 450 mg (Starting Dose in TIW Dosing Regimen) | Vadadustat 600 mg (Starting Dose in TIW Dosing Regimen) | Vadadustat 750 mg (Starting Dose in TIW Dosing Regimen) | Vadadustat Total (TIW Dosing Regimen) | ESA Hyporesponder Parallel Study: Vadadustat ≤ 750 mg (TIW Dosing Regimen)
Number analyzed (Participants) | 1 | 4 | 7 | 5 | 17 | 0
g/dL | -0.050 (NA) — Standard deviation cannot be calculated due to only one participant with data | -1.021 (1.0961) | -0.360 (0.4894) | -0.103 (1.9225) | -0.422 (1.1708) |

8. Secondary Outcome: Mean Change in Hb Between Baseline and the SEP
Description: Change from Baseline was calculated as the SEP value minus the Baseline value. The Baseline Hb value was defined as the average of the final two Hb values prior to start of dosing on Day 1. The SEP value was the average Hb value from Week 18 to Week 20.
Time Frame: Baseline; Week 18 to Week 20
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Low Dose of Epoetin Alfa: Vadadustat 300 mg | Low Dose of Epoetin Alfa: Vadadustat 450 mg | Low Dose of Epoetin Alfa: Epoetin Alfa | High Dose of Epoetin Alfa: Vadadustat 300 mg | High Dose of Epoetin Alfa: Vadadustat 450 mg | High Dose of Epoetin Alfa: Vadadustat 600 mg | High Dose of Epoetin Alfa: Epoetin Alfa | ESA Hyporesponder: Vadadustat 600 mg | ESA Hyporesponder: Epoetin Alfa
Number analyzed (Participants) | 26 | 24 | 23 | 7 | 14 | 10 | 12 | 3 | 4
g/dL | -0.197 (1.1597) | -0.186 (0.8703) | 0.070 (0.9545) | 0.114 (1.0242) | -0.421 (0.8370) | -0.545 (0.9771) | 0.343 (0.8897) | -0.283 (0.7371) | -0.400 (1.0157)

9. Secondary Outcome: Number of Participants With Hb Values Within the Target Range at the SEP
Description: The target range for Hb was from 10.0 to 11.0 g/dL. The SEP was comprised of Week 18 to Week 20.
Time Frame: Week 18 to Week 20
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose of Epoetin Alfa: Vadadustat 300 mg | Low Dose of Epoetin Alfa: Vadadustat 450 mg | Low Dose of Epoetin Alfa: Epoetin Alfa | High Dose of Epoetin Alfa: Vadadustat 300 mg | High Dose of Epoetin Alfa: Vadadustat 450 mg | High Dose of Epoetin Alfa: Vadadustat 600 mg | High Dose of Epoetin Alfa: Epoetin Alfa | ESA Hyporesponder: Vadadustat 600 mg | ESA Hyporesponder: Epoetin Alfa
Number analyzed (Participants) | 26 | 24 | 23 | 7 | 14 | 10 | 12 | 3 | 4
Participants | 6 | 7 | 9 | 2 | 3 | 2 | 6 | 1 | 1

10. Secondary Outcome: Number of Participants With Hb Values Within the Target Range at the SEP in Participants Who Transitioned to TIW Vadadustat Dosing
Description: The target range for Hb was from 10.0 to 11.0 g/dL. The SEP was comprised of Week 18 to Week 20. For the Main Study, analysis is presented per dose level according to the starting dose in TIW regimen, as well as being presented as a combined arm for "Vadadustat Total (TIW dosing regimen)". For the ESA Hyporesponder Parallel Study, a starting dose classification for TIW dosing regimen was not applicable due to no participants switching from Vadadustat QD to TIW dosing.
Time Frame: Week 18 to Week 20
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Groups:
- ESA Hyporesponder Parallel Study: Vadadustat ≤ 750 mg (TIW Dosing Regimen): After completing the 12-week QD dosing regimen, eligible participants based on investigator's discretion were switched from daily dosing to TIW dosing to receive a starting dose of Vadadustat ≤ 750 mg (1 tablet greater [150 mg] than final dose in QD dosing regimen. Participants who reported a decline in Hb ≥0.5 g/dL were eligible for a dose increase by another 150 mg until Week 20.
Arm/Group | Vadadustat 300 mg (Starting Dose in TIW Dosing Regimen) | Vadadustat 450 mg (Starting Dose in TIW Dosing Regimen) | Vadadustat 600 mg (Starting Dose in TIW Dosing Regimen) | Vadadustat 750 mg (Starting Dose in TIW Dosing Regimen) | Vadadustat Total (TIW Dosing Regimen) | ESA Hyporesponder Parallel Study: Vadadustat ≤ 750 mg (TIW Dosing Regimen)
Number analyzed (Participants) | 1 | 4 | 7 | 5 | 17 | 0
Participants | 0 | 2 | 2 | 3 | 7 |

11. Secondary Outcome: Number of Participants With a Mean Increase in Hb From Baseline to the PEP ≥0.5 g/dL or With Hb Values Within the Target Range at the PEP
Description: The target range for Hb was from 10.0 to 11.0 g/dL. The PEP was comprised of Week 10 to Week 12.
Time Frame: Week 10 to Week 12
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose of Epoetin Alfa: Vadadustat 300 mg | Low Dose of Epoetin Alfa: Vadadustat 450 mg | Low Dose of Epoetin Alfa: Epoetin Alfa | High Dose of Epoetin Alfa: Vadadustat 300 mg | High Dose of Epoetin Alfa: Vadadustat 450 mg | High Dose of Epoetin Alfa: Vadadustat 600 mg | High Dose of Epoetin Alfa: Epoetin Alfa | ESA Hyporesponder: Vadadustat 600 mg | ESA Hyporesponder: Epoetin Alfa
Number analyzed (Participants) | 30 | 30 | 23 | 12 | 18 | 14 | 12 | 4 | 5
Participants | 14 | 19 | 18 | 1 | 6 | 6 | 8 | 0 | 1

12. Secondary Outcome: Number of Participants With a Mean Increase in Hb From Baseline to the SEP ≥0.5 g/dL or With Hb Values Within the Target Range at the SEP
Description: The target range for Hb was from 10.0 to 11.0 grams per g/dL. The SEP was comprised of Week 18 to Week 20.
Time Frame: Week 18 to Week 20
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Groups:
- Stratum 1 (Epoetin Alfa ≤90 U/kg/Week): Vadadustat 300 mg: Participants who were maintained on the low dose of Epoetin Alfa (≤90 units per kilogram per week [U/kg/week]) prior to and including the Screening Period for a minimum of 8 weeks prior to Screening Visit 2 were administered an oral dose of Vadadustat 300 milligram (mg) tablet per day (QD) until Week 12. Eligible participants based on investigator's discretion were switched from daily dosing to three times per week (TIW) dosing of the starting Vadadustat dose (300 mg) plus a 150 mg greater dose (450 mg) to maintain target hemoglobin (Hb) levels during Week 12 to Week 14. Non-eligile participants continued with daily dosing. Participants who reported a decline in Hb ≥0.5 grams per deciliter (g/dL) were eligible for a dose increase by another 150 mg until Week 20.
- Stratum 1 (Epoetin Alfa ≤90 U/kg/Week): Vadadustat 450 mg: Participants who were maintained on the low dose of Epoetin Alfa (≤90 U/kg/week) prior to and including the Screening Period for a minimum of 8 weeks prior to Screening Visit 2 were administered an oral dose of Vadadustat 450 mg tablet QD until Week 12. Eligible participants based on investigator's discretion were switched from daily dosing to TIW dosing of the starting Vadadustat dose (450 mg) plus a 150 mg greater dose (600 mg) to maintain target Hb levels during Week 12 to Week 14. Non-eligible participants continued with daily dosing. Participants who reported a decline in Hb ≥0.5 g/dL were eligible for a dose increase by another 150 mg until Week 20.
- Stratum 1 (Epoetin Alfa ≤90 U/kg/Week): Epoetin Alfa: Participants who were maintained on the low dose of Epoetin Alfa (≤90 U/kg/week) prior to and including the screening period for a minimum of 8 weeks prior to screening visit 2, were administered with three times a week (TIW) dose of Epoetin Alfa based on the participant's central laboratory hemoglobin (Hb) value and the approved Epoetin Alfa United States (US) Package Insert (PI) for adult participants with CKD on dialysis. Dose was adjusted to achieve and maintain Hb levels within the target range of 10.0 and 11.0 g/dL, inclusive.
- ESA Hyporesponder (Epoetin Alfa ≥300 U/kg/Week): Vadadustat 600 mg: In the erythropoiesis-stimulating agent (ESA) hyporesponder parallel study participants who were maintained on ≥300 U/kg/week dose of Epoetin Alfa prior to and including the screening period for a minimum of 8 weeks prior to screening visit 2, were administered with an oral dose of Vadadustat 600 mg tablet per day.
- ESA Hyporesponder (Epoetin Alfa ≥300 U/kg/Week): Epoetin Alfa: In the ESA hyporesponder parallel study participants who were maintained on ≥300 U/kg/week dose of Epoetin Alfa prior to and including the screening period for a minimum of 8 weeks prior to screening visit 2, were administered with three TIW dose of Epoetin Alfa based on the participant's central laboratory Hb value and the approved Epoetin Alfa US PI for adult participants with CKD on dialysis. Dose was adjusted to achieve and maintain Hb levels within the target range of 10.0 and 11.0 g/dL, inclusive.
Arm/Group | Stratum 1 (Epoetin Alfa ≤90 U/kg/Week): Vadadustat 300 mg | Stratum 1 (Epoetin Alfa ≤90 U/kg/Week): Vadadustat 450 mg | Stratum 1 (Epoetin Alfa ≤90 U/kg/Week): Epoetin Alfa | High Dose of Epoetin Alfa: Vadadustat 300 mg | High Dose of Epoetin Alfa: Vadadustat 450 mg | High Dose of Epoetin Alfa: Vadadustat 600 mg | High Dose of Epoetin Alfa: Epoetin Alfa | ESA Hyporesponder (Epoetin Alfa ≥300 U/kg/Week): Vadadustat 600 mg | ESA Hyporesponder (Epoetin Alfa ≥300 U/kg/Week): Epoetin Alfa
Number analyzed (Participants) | 26 | 24 | 23 | 7 | 14 | 10 | 12 | 3 | 4
Participants | 10 | 11 | 14 | 3 | 5 | 2 | 8 | 1 | 2

13. Secondary Outcome: Number of Participants Requiring at Least One Intravenous (IV) Elemental Iron Supplementation
Description: Iron supplementation was performed to maintain ferritin ≥200 nanograms/milliliters (ng/mL) and transferrin saturation (TSAT) ≥20%.
Time Frame: Up to Week 20
Population: Randomized Population. Analysis of this population was based on the randomized treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose of Epoetin Alfa: Vadadustat 300 mg | Low Dose of Epoetin Alfa: Vadadustat 450 mg | Low Dose of Epoetin Alfa: Epoetin Alfa | High Dose of Epoetin Alfa: Vadadustat 300 mg | High Dose of Epoetin Alfa: Vadadustat 450 mg | High Dose of Epoetin Alfa: Vadadustat 600 mg | High Dose of Epoetin Alfa: Epoetin Alfa | ESA Hyporesponder: Vadadustat 600 mg | ESA Hyporesponder: Epoetin Alfa
Number analyzed (Participants) | 35 | 34 | 23 | 18 | 21 | 21 | 13 | 5 | 5
Participants | 23 | 21 | 16 | 10 | 14 | 18 | 10 | 4 | 5

14. Secondary Outcome: Number of Participants Requiring Erythropoiesis-stimulating Agent (ESA) Rescue
Description: ESA rescue therapy was administered in participants with Hb ≥8.5 g/dL, and was stopped when Hb reached ≥9.0 g/dL.
Time Frame: Up to Week 20
Population: Randomized Population. Analysis of this population was based on the randomized treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose of Epoetin Alfa: Vadadustat 300 mg | Low Dose of Epoetin Alfa: Vadadustat 450 mg | Low Dose of Epoetin Alfa: Epoetin Alfa | High Dose of Epoetin Alfa: Vadadustat 300 mg | High Dose of Epoetin Alfa: Vadadustat 450 mg | High Dose of Epoetin Alfa: Vadadustat 600 mg | High Dose of Epoetin Alfa: Epoetin Alfa | ESA Hyporesponder: Vadadustat 600 mg | ESA Hyporesponder: Epoetin Alfa
Number analyzed (Participants) | 35 | 34 | 23 | 18 | 21 | 21 | 13 | 5 | 5
Participants | 2 | 8 | 3 | 5 | 5 | 3 | 1 | 3 | 1

15. Secondary Outcome: Number of Participants Requiring Red Blood Cell (RBC) Transfusion
Description: RBC transfusion was administered as rescue therapy in the event of an acute or severe loss of blood.
Time Frame: Up to Week 20
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose of Epoetin Alfa: Vadadustat 300 mg | Low Dose of Epoetin Alfa: Vadadustat 450 mg | Low Dose of Epoetin Alfa: Epoetin Alfa | High Dose of Epoetin Alfa: Vadadustat 300 mg | High Dose of Epoetin Alfa: Vadadustat 450 mg | High Dose of Epoetin Alfa: Vadadustat 600 mg | High Dose of Epoetin Alfa: Epoetin Alfa | ESA Hyporesponder: Vadadustat 600 mg | ESA Hyporesponder: Epoetin Alfa
Number analyzed (Participants) | 35 | 34 | 23 | 18 | 21 | 21 | 13 | 5 | 5
Participants | 0 | 1 | 0 | 3 | 1 | 2 | 0 | 1 | 1

16. Secondary Outcome: Mean Serum Concentration of Erythropoietin (EPO) for Vadadustat Treatment Groups by Strata of Epoetin Alfa Dose Group
Description: Blood samples were collected from participants at defined time points for the assessment of EPO concentration. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline; Week 1 (pre-dose), Week 1 +1 (Day 8; pre-dose), Week 11 (pre-dose), and Week 13 (pre-dose)
Population: Pharmacokinetic (PK) Population: all randomized participants who received study drug and had enough drug concentrations to estimate AUC and Cmax. Analysis of this population was based on the dose amount taken at the date of PK sampling for the Vadadustat group. Participants with concentrations below the limit of quantitation (BLQ) for all the time points were excluded from the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Milliunits per milliliter
Arm/Group | Low Dose of Epoetin Alfa: Vadadustat 300 mg | Low Dose of Epoetin Alfa: Vadadustat 450 mg | High Dose of Epoetin Alfa: Vadadustat 300 mg | High Dose of Epoetin Alfa: Vadadustat 450 mg | High Dose of Epoetin Alfa: Vadadustat 600 mg | ESA Hyporesponder: Vadadustat 600 mg
Number analyzed (Participants) | 33 | 30 | 15 | 21 | 15 | 5
Milliunits per milliliter
  Baseline: number analyzed (Participants) | 33 | 30 | 12 | 17 | 14 | 5
  Baseline | 7.33 (57.3) | 9.53 (54.0) | 9.93 (83.6) | 8.77 (48.2) | 6.98 (61.6) | 8.03 (53.2)
  Week 1: number analyzed (Participants) | 33 | 27 | 15 | 20 | 15 | 5
  Week 1 | 12.1 (94.3) | 17.5 (97.0) | 15.3 (72.6) | 14.1 (86.4) | 20.2 (90.8) | 12.9 (54.2)
  Week 1 +1 (Day 8): number analyzed (Participants) | 30 | 27 | 13 | 21 | 12 | 5
  Week 1 +1 (Day 8) | 15.6 (76.3) | 18.9 (98.2) | 16.1 (76.0) | 18.0 (49.8) | 17.4 (104.8) | 9.49 (37.1)
  Week 11: number analyzed (Participants) | 12 | 15 | 4 | 4 | 8 | 0
  Week 11 | 14.2 (55.9) | 14.9 (106.2) | 19.4 (78.0) | 20.6 (169.6) | 17.3 (53.4) |
  Week 13: number analyzed (Participants) | 0 | 4 | 1 | 0 | 2 | 0
  Week 13 |  | 15.7 (107.2) | 39.2 (NA) — Dispersion data are not available for a single participant. |  | 10.5 (47.1) |

17. Secondary Outcome: Mean Change From Baseline in Reticulocyte Count
Description: Blood samples were collected from participants at defined time points for the assessment of reticulocyte count. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline; Week 1, Week 4, Week 8, Week 11, Week 12, Week 13, Week 16, and Week 20
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: 10^3 cells/microliter (µL)
Arm/Group | Low Dose of Epoetin Alfa: Vadadustat 300 mg | Low Dose of Epoetin Alfa: Vadadustat 450 mg | Low Dose of Epoetin Alfa: Epoetin Alfa | High Dose of Epoetin Alfa: Vadadustat 300 mg | High Dose of Epoetin Alfa: Vadadustat 450 mg | High Dose of Epoetin Alfa: Vadadustat 600 mg | High Dose of Epoetin Alfa: Epoetin Alfa | ESA Hyporesponder: Vadadustat 600 mg | ESA Hyporesponder: Epoetin Alfa
Number analyzed (Participants) | 30 | 32 | 21 | 18 | 20 | 21 | 11 | 5 | 5
10^3 cells/microliter (µL)
  Baseline | 51.9 (27.57) | 47.2 (17.81) | 48.8 (27.27) | 59.3 (42.02) | 48.4 (33.45) | 51.5 (25.14) | 62.6 (25.88) | 77.6 (51.04) | 83.0 (45.34)
  Week 1: number analyzed (Participants) | 23 | 21 | 16 | 11 | 16 | 16 | 10 | 5 | 5
  Week 1 | 3.1 (24.09) | 6.9 (30.60) | 1.0 (22.42) | -18.1 (24.81) | -3.9 (28.51) | -6.6 (33.80) | 20.4 (48.64) | -35.8 (45.06) | -25.2 (29.73)
  Week 4: number analyzed (Participants) | 25 | 25 | 17 | 15 | 19 | 15 | 11 | 5 | 5
  Week 4 | 14.6 (32.25) | 14.9 (29.45) | 0.8 (40.68) | -5.6 (37.38) | 2.9 (39.68) | 6.1 (33.24) | 22.5 (50.53) | -26.8 (55.44) | 17.5 (26.21)
  Week 8: number analyzed (Participants) | 22 | 24 | 18 | 12 | 14 | 11 | 8 | 4 | 5
  Week 8 | 14.0 (31.40) | 23.9 (39.26) | 23.1 (38.98) | 9.1 (46.38) | 20.4 (49.42) | 23.1 (20.33) | 14.0 (54.60) | -3.3 (67.56) | -21.8 (69.36)
  Week 11: number analyzed (Participants) | 21 | 19 | 17 | 9 | 15 | 9 | 9 | 3 | 5
  Week 11 | 11.7 (25.06) | 20.2 (25.80) | 21.0 (35.12) | 26.2 (26.2) | 32.5 (70.42) | 9.2 (41.30) | 3.9 (46.15) | -6.7 (76.89) | -27.2 (71.36)
  Week 12: number analyzed (Participants) | 20 | 21 | 18 | 7 | 14 | 11 | 9 | 4 | 4
  Week 12 | 16.1 (32.60) | 16.3 (34.27) | 22.2 (26.72) | 47.7 (66.66) | 20.3 (44.30) | 26.9 (52.64) | 4.6 (39.53) | 3.8 (52.72) | -17.3 (67.06)
  Week 13: number analyzed (Participants) | 22 | 20 | 17 | 6 | 12 | 8 | 10 | 2 | 3
  Week 13 | 16.7 (27.07) | 12.1 (43.12) | 16.4 (26.53) | 46.3 (57.25) | 15.9 (43.79) | 10.5 (28.80) | 0.1 (46.05) | 2.0 (83.44) | 16.3 (11.93)
  Week 16: number analyzed (Participants) | 21 | 21 | 19 | 5 | 9 | 10 | 7 | 2 | 4
  Week 16 | 13.9 (35.40) | 19.6 (37.61) | 8.3 (34.16) | -2.2 (57.32) | 9.7 (30.17) | 0.2 (22.08) | 26.6 (55.82) | -31.5 (86.97) | 4.0 (16.21)
  Week 20: number analyzed (Participants) | 20 | 16 | 19 | 7 | 12 | 8 | 10 | 3 | 2
  Week 20 | 14.5 (25.74) | 13.2 (24.50) | 23.8 (26.49) | 10.3 (41.33) | 16.4 (35.54) | 10.9 (29.81) | 38.5 (44.11) | -3.3 (52.58) | 40.0 (7.07)

18. Secondary Outcome: Mean Change From Baseline in Iron Concentration
Description: Blood samples were collected from participants at defined time points for the assessment of iron indices, including iron concentration. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline; Week 4, Week 8, Week 12, Week 16, and Week 20
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: micrograms per deciliter (µg/dL)
Arm/Group | Low Dose of Epoetin Alfa: Vadadustat 300 mg | Low Dose of Epoetin Alfa: Vadadustat 450 mg | Low Dose of Epoetin Alfa: Epoetin Alfa | High Dose of Epoetin Alfa: Vadadustat 300 mg | High Dose of Epoetin Alfa: Vadadustat 450 mg | High Dose of Epoetin Alfa: Vadadustat 600 mg | High Dose of Epoetin Alfa: Epoetin Alfa | ESA Hyporesponder: Vadadustat 600 mg | ESA Hyporesponder: Epoetin Alfa
Number analyzed (Participants) | 35 | 34 | 23 | 18 | 21 | 21 | 13 | 5 | 5
micrograms per deciliter (µg/dL)
  Baseline | 87.4 (38.46) | 93.9 (36.56) | 90.1 (35.09) | 57.7 (26.71) | 80.9 (36.94) | 73.1 (22.23) | 65.7 (23.93) | 81.6 (37.01) | 58.4 (18.77)
  Week 4: number analyzed (Participants) | 31 | 29 | 20 | 16 | 20 | 15 | 13 | 5 | 4
  Week 4 | -8.0 (34.49) | -11.2 (33.59) | -18.3 (22.83) | 3.3 (35.23) | 9.6 (29.67) | 1.7 (23.37) | -6.6 (32.86) | 8.6 (17.36) | 3.8 (25.79)
  Week 8: number analyzed (Participants) | 31 | 27 | 21 | 12 | 17 | 12 | 11 | 4 | 5
  Week 8 | -5.5 (45.04) | -15.0 (40.51) | -8.6 (44.30) | 4.5 (24.06) | -5.9 (36.91) | 11.7 (40.33) | -12.6 (26.55) | 0.3 (11.09) | 2.0 (20.33)
  Week 12: number analyzed (Participants) | 24 | 25 | 18 | 8 | 14 | 10 | 9 | 4 | 5
  Week 12 | -2.7 (38.24) | -22.2 (43.14) | -26.0 (33.03) | -2.8 (40.49) | -0.4 (40.20) | -5.1 (27.54) | -16.1 (22.88) | -2.5 (43.94) | -12.6 (28.99)
  Week 16: number analyzed (Participants) | 26 | 24 | 21 | 7 | 10 | 10 | 10 | 2 | 4
  Week 16 | -22.8 (39.39) | -18.3 (39.85) | -17.9 (53.89) | -0.7 (10.26) | 5.2 (30.27) | -4.6 (30.31) | -13.9 (44.05) | 19.5 (53.03) | -12.0 (24.06)
  Week 20: number analyzed (Participants) | 26 | 23 | 21 | 7 | 13 | 8 | 12 | 3 | 3
  Week 20 | -14.2 (41.11) | -9.5 (27.87) | -16.6 (46.49) | 28.7 (67.73) | -3.1 (32.43) | 13.4 (16.03) | -8.4 (28.94) | -15.3 (43.19) | -10.3 (21.57)

19. Secondary Outcome: Mean Change From Baseline in Ferritin Concentration
Description: Blood samples were collected from participants at defined time points for the assessment of iron indices, including ferritin concentration. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline; Week 4, Week 8, Week 12, Week 16, and Week 20
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: micrograms per liter (µg/L)
Arm/Group | Low Dose of Epoetin Alfa: Vadadustat 300 mg | Low Dose of Epoetin Alfa: Vadadustat 450 mg | Low Dose of Epoetin Alfa: Epoetin Alfa | High Dose of Epoetin Alfa: Vadadustat 300 mg | High Dose of Epoetin Alfa: Vadadustat 450 mg | High Dose of Epoetin Alfa: Vadadustat 600 mg | High Dose of Epoetin Alfa: Epoetin Alfa | ESA Hyporesponder: Vadadustat 600 mg | ESA Hyporesponder: Epoetin Alfa
Number analyzed (Participants) | 34 | 34 | 23 | 18 | 21 | 21 | 13 | 5 | 5
micrograms per liter (µg/L)
  Baseline | 939.3 (478.64) | 1043.6 (359.10) | 919.3 (298.27) | 910.2 (408.03) | 745.2 (362.98) | 739.5 (329.66) | 723.6 (484.29) | 1182.2 (508.67) | 449.6 (423.44)
  Week 4: number analyzed (Participants) | 31 | 29 | 20 | 16 | 20 | 15 | 13 | 5 | 4
  Week 4 | -30.1 (185.45) | -101.9 (204.51) | -23.7 (274.39) | 41.4 (335.00) | 152.9 (347.97) | 45.5 (320.50) | -145.6 (211.10) | 34.8 (470.43) | -61.5 (17.37)
  Week 8: number analyzed (Participants) | 31 | 26 | 21 | 12 | 17 | 12 | 11 | 4 | 5
  Week 8 | -120.8 (273.28) | -185.4 (298.19) | 24.9 (334.28) | 29.4 (361.29) | -5.6 (255.10) | -87.8 (285.30) | -78.3 (254.98) | 111.3 (609.61) | 397.8 (453.76)
  Week 12: number analyzed (Participants) | 24 | 25 | 17 | 8 | 14 | 10 | 9 | 4 | 5
  Week 12 | -118.5 (220.40) | -194.8 (288.47) | -42.4 (356.19) | -68.0 (275.11) | -23.8 (303.39) | -30.1 (386.24) | -195.3 (304.63) | -0.5 (237.99) | -35.0 (157.46)
  Week 16: number analyzed (Participants) | 26 | 24 | 21 | 7 | 10 | 10 | 10 | 2 | 4
  Week 16 | -92.0 (309.88) | -70.9 (288.34) | 99.5 (567.19) | -144.0 (358.78) | 27.8 (244.67) | -97.2 (188.15) | -81.8 (447.01) | 80.0 (243.24) | 62.3 (186.15)
  Week 20: number analyzed (Participants) | 26 | 23 | 21 | 7 | 13 | 8 | 12 | 3 | 3
  Week 20 | -113.6 (327.06) | -166.6 (298.67) | 26.5 (497.52) | -199.4 (370.32) | 4.8 (331.76) | -51.6 (253.07) | -104.8 (347.53) | 249.0 (636.33) | 607.0 (607.0)

20. Secondary Outcome: Mean Change From Baseline in Total Iron Binding Capacity
Description: Blood samples were collected from participants at defined time points for the assessment of iron indices, including Total Iron Binding Capacity. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline; Week 4, Week 8, Week 12, Week 16, and Week 20
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: µg/dL
Arm/Group | Low Dose of Epoetin Alfa: Vadadustat 300 mg | Low Dose of Epoetin Alfa: Vadadustat 450 mg | Low Dose of Epoetin Alfa: Epoetin Alfa | High Dose of Epoetin Alfa: Vadadustat 300 mg | High Dose of Epoetin Alfa: Vadadustat 450 mg | High Dose of Epoetin Alfa: Vadadustat 600 mg | High Dose of Epoetin Alfa: Epoetin Alfa | ESA Hyporesponder: Vadadustat 600 mg | ESA Hyporesponder: Epoetin Alfa
Number analyzed (Participants) | 35 | 34 | 23 | 18 | 21 | 21 | 13 | 5 | 5
µg/dL
  Baseline | 237.8 (39.28) | 230.7 (39.09) | 234.8 (44.76) | 210.1 (33.33) | 235.7 (38.80) | 223.6 (34.31) | 218.2 (33.80) | 211.0 (42.99) | 225.6 (98.15)
  Week 4: number analyzed (Participants) | 31 | 29 | 20 | 16 | 20 | 15 | 13 | 5 | 4
  Week 4 | 35.9 (27.11) | 27.7 (33.58) | -13.4 (26.02) | 27.6 (28.49) | 41.0 (26.22) | 48.2 (37.78) | -0.5 (21.44) | 44.2 (53.58) | 7.8 (14.38)
  Week 8: number analyzed (Participants) | 31 | 27 | 21 | 12 | 17 | 12 | 11 | 4 | 5
  Week 8 | 30.3 (28.42) | 37.0 (40.99) | -1.1 (18.38) | 26.3 (23.98) | 49.4 (27.34) | 58.8 (24.54) | -7.4 (19.26) | 56.0 (58.15) | -24.8 (58.79)
  Week 12: number analyzed (Participants) | 24 | 25 | 18 | 8 | 14 | 10 | 9 | 4 | 5
  Week 12 | 42.4 (27.10) | 37.2 (43.09) | -9.9 (25.85) | 25.1 (33.90) | 41.0 (39.05) | 54.5 (44.05) | -3.8 (25.42) | 58.0 (14.45) | -0.6 (15.32)
  Week 16: number analyzed (Participants) | 26 | 24 | 21 | 7 | 10 | 10 | 10 | 2 | 4
  Week 16 | 35.0 (43.00) | 27.8 (35.16) | -3.0 (25.44) | 55.3 (28.63) | 53.1 (58.33) | 60.9 (70.50) | -13.7 (31.46) | 42.5 (62.93) | -2.5 (18.52)
  Week 20: number analyzed (Participants) | 26 | 23 | 21 | 7 | 13 | 8 | 12 | 3 | 3
  Week 20 | 38.0 (28.15) | 44.9 (30.71) | -9.5 (29.29) | 51.7 (37.50) | 68.4 (43.40) | 67.9 (58.44) | -5.4 (29.78) | 66.7 (35.22) | -6.0 (21.79)

21. Secondary Outcome: Mean Change From Baseline in Hepcidin Concentration
Description: Blood samples were collected from participants at defined time points for the assessment of hepcidin concentration. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline; Week 12 and Week 20
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Groups:
- ESA Hyporesponder: Epoetin Alfa: In the ESA hyporesponder parallel study participants who were maintained on ≥300 U/kg/week dose of Epoetin Alfa prior to and including the screening period for a minimum of 8 weeks prior to screening visit 2, were administered with three TIW dose of Epoetin Alfa based on the participant's central laboratory Hb value and the approved Epoetin Alfa US PI for adult participants with CKD on dialysis. Dose was adjusted to achieve and maintain Hb levels within the target range of 10.0 and 11.0 g/dL, inclusive.(US) Package Insert (PI) for adult participants with CKD on dialysis. Dose was adjusted to achieve and maintain Hb levels within the target range of 10.0 and 11.0 g/dL, inclusive"
Arm/Group | Low Dose of Epoetin Alfa: Vadadustat 300 mg | Low Dose of Epoetin Alfa: Vadadustat 450 mg | Low Dose of Epoetin Alfa: Epoetin Alfa | High Dose of Epoetin Alfa: Vadadustat 300 mg | High Dose of Epoetin Alfa: Vadadustat 450 mg | High Dose of Epoetin Alfa: Vadadustat 600 mg | High Dose of Epoetin Alfa: Epoetin Alfa | ESA Hyporesponder: Vadadustat 600 mg | ESA Hyporesponder: Epoetin Alfa
Number analyzed (Participants) | 35 | 34 | 21 | 17 | 21 | 21 | 13 | 5 | 5
nanograms per milliliter (ng/mL)
  Baseline | 194.870 (113.9348) | 208.816 (85.1667) | 259.161 (134.9995) | 185.852 (105.6611) | 215.608 (130.7350) | 160.760 (102.6261) | 143.519 (124.6749) | 239.958 (151.3859) | 74.748 (40.2119)
  Week 12: number analyzed (Participants) | 24 | 24 | 17 | 7 | 14 | 10 | 9 | 3 | 5
  Week 12 | -50.565 (57.6474) | -53.675 (92.1185) | -66.646 (152.3178) | -55.283 (77.1648) | -34.868 (89.7176) | -74.797 (126.1667) | -62.787 (96.1842) | -128.587 (262.6300) | -1.062 (30.4842)
  Week 20: number analyzed (Participants) | 24 | 23 | 17 | 6 | 13 | 8 | 10 | 3 | 3
  Week 20 | -86.025 (100.4382) | -38.627 (75.0555) | -83.685 (95.7049) | -93.412 (115.2839) | -83.012 (98.7521) | -43.701 (80.8411) | -80.680 (125.2481) | -152.243 (218.9284) | -9.023 (80.4001)

22. Secondary Outcome: Geometric Mean Maximum Observed Plasma Concentration (Cmax) of Vadadustat Following a Single Dose
Description: Blood samples were collected from participants at defined time points for the assessment of Cmax of Vadadustat following a single dose.
Time Frame: Day 1; Week 1, Week 1 +1 (Day 8), Week 11, Week 13: pre-dose, 2 hours (h), 3.5h, and 5h post-dose, and additionally at 7h and 10.5h post-dose
Population: PK Population. Analysis of this population was based on the dose amount taken at the date of PK sampling for the Vadadustat group. Participants with non-missing values were included in the analysis. PK parameter of plasma Vadadustat concentration for Vadadustat treatment groups without dose normalization by strata of Epoetin Alfa dose group were included for the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter (μg/mL)
Arm/Group | Low Dose of Epoetin Alfa: Vadadustat 300 mg | Low Dose of Epoetin Alfa: Vadadustat 450 mg | High Dose of Epoetin Alfa: Vadadustat 300 mg | High Dose of Epoetin Alfa: Vadadustat 450 mg | High Dose of Epoetin Alfa: Vadadustat 600 mg | ESA Hyporesponder: Vadadustat 600 mg
Number analyzed (Participants) | 32 | 30 | 14 | 21 | 17 | 5
Micrograms per milliliter (μg/mL)
  Week 1 | 26.0 (87.9) | 40.8 (54.8) | 26.5 (59.3) | 47.0 (38.2) | 56.5 (39.2) | 44.2 (73.1)
  Week 1 +1 (Day 8): number analyzed (Participants) | 30 | 30 | 14 | 21 | 13 | 5
  Week 1 +1 (Day 8) | 20.1 (174.4) | 37.6 (78.9) | 23.8 (69.0) | 44.2 (29.6) | 60.1 (41.6) | 31.6 (151.6)
  Week 11: number analyzed (Participants) | 12 | 15 | 5 | 4 | 8 | 0
  Week 11 | 28.6 (49.3) | 24.4 (350.6) | 32.4 (26.9) | 38.1 (99.0) | 41.2 (77.7) |
  Week 13: number analyzed (Participants) | 0 | 4 | 1 | 0 | 2 | 0
  Week 13 |  | 30.6 (102.7) | 11.5 (NA) — Dispersion data are not available for a single participant |  | 60.2 (9.2) |

23. Secondary Outcome: Geometric Mean Area Under the Concentration-time Curve (AUC) From Time 0 to 24 Hours (AUC0-24) of Vadadustat Following a Single Dose
Description: Blood samples were collected from participants at defined time points for the assessment of AUC and AUC0-24 of Vadadustat following a single dose.
Time Frame: Day 1; Week 1, Week 1 +1 (Day 8), Week 11: pre-dose, 2h, 3.5h, and 5h post-dose, and additionally at 7h and 10.5h post-dose
Population: as for outcome 22
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*µg/mL
Arm/Group | Low Dose of Epoetin Alfa: Vadadustat 300 mg | Low Dose of Epoetin Alfa: Vadadustat 450 mg | High Dose of Epoetin Alfa: Vadadustat 300 mg | High Dose of Epoetin Alfa: Vadadustat 450 mg | High Dose of Epoetin Alfa: Vadadustat 600 mg | ESA Hyporesponder: Vadadustat 600 mg
Number analyzed (Participants) | 29 | 28 | 13 | 21 | 13 | 5
hours*µg/mL
  Week 1: number analyzed (Participants) | 27 | 23 | 11 | 19 | 12 | 5
  Week 1 | 338 (63.8) | 518 (71.1) | 342 (81.7) | 605 (54.5) | 786 (36.6) | 464 (80.9)
  Week 1 +1 (Day 8) | 289 (76.6) | 465 (80.8) | 310 (94.7) | 566 (41.1) | 847 (54.8) | 388 (112.4)
  Week 11: number analyzed (Participants) | 11 | 14 | 5 | 4 | 8 | 0
  Week 11 | 344 (53.5) | 338 (282.0) | 402 (70.8) | 450 (68.2) | 588 (52.5) |

24. Secondary Outcome: Median Terminal Half-life (t1/2) of Vadadustat Following a Single Dose
Description: Blood samples were collected from participants at defined time points for the assessment of t1/2 of Vadadustat following a single dose.
Time Frame: as for outcome 22
Population: as for outcome 22
Measure: Median (Full Range); unit: Hours
Arm/Group | Low Dose of Epoetin Alfa: Vadadustat 300 mg | Low Dose of Epoetin Alfa: Vadadustat 450 mg | High Dose of Epoetin Alfa: Vadadustat 300 mg | High Dose of Epoetin Alfa: Vadadustat 450 mg | High Dose of Epoetin Alfa: Vadadustat 600 mg | ESA Hyporesponder: Vadadustat 600 mg
Number analyzed (Participants) | 17 | 17 | 8 | 8 | 6 | 2
Hours
  Week 1: number analyzed (Participants) | 17 | 17 | 7 | 8 | 5 | 2
  Week 1 | 8.53 [5.36 to 26.6] | 10.5 [3.26 to 21.1] | 12.5 [7.33 to 20.7] | 10.3 [6.33 to 18.3] | 11.0 [6.51 to 18.0] | 9.01 [8.45 to 9.58]
  Week 1 +1 (Day 8): number analyzed (Participants) | 13 | 16 | 8 | 8 | 6 | 2
  Week 1 +1 (Day 8) | 8.82 [5.80 to 22.9] | 8.83 [4.98 to 70.0] | 10.1 [4.79 to 17.9] | 12.4 [5.73 to 47.8] | 14.6 [5.61 to 31.3] | 11.7 [11.3 to 12.0]
  Week 11: number analyzed (Participants) | 6 | 6 | 2 | 1 | 3 | 0
  Week 11 | 6.73 [3.55 to 22.1] | 10.4 [6.46 to 13.8] | 6.49 [3.22 to 9.75] | 3.95 [3.95 to 3.95] | 5.65 [5.26 to 7.12] |
  Week 13: number analyzed (Participants) | 0 | 1 | 0 | 0 | 1 | 0
  Week 13 |  | 11.0 [11.0 to 11.0] |  |  | 5.01 [5.01 to 5.01] |

25. Secondary Outcome: Median Time to Reach Cmax (Tmax) of Vadadustat Following a Single Dose
Description: Blood samples were collected from participants at defined time points for the assessment of Tmax of Vadadustat following a single dose.
Time Frame: as for outcome 22
Population: PK Population. Analysis of this population was based on the dose amount taken at the date of PK sampling for Vadadustat group. Participants with non-missing values were included in the analysis. PK parameter of plasma Vadadustat concentration for Vadadustat treatment groups without dose normalization by strata of Epoetin Alfa dose group were included for the analysis.
Measure: Median (Full Range); unit: Hours
Arm/Group | Low Dose of Epoetin Alfa: Vadadustat 300 mg | Low Dose of Epoetin Alfa: Vadadustat 450 mg | High Dose of Epoetin Alfa: Vadadustat 300 mg | High Dose of Epoetin Alfa: Vadadustat 450 mg | High Dose of Epoetin Alfa: Vadadustat 600 mg | ESA Hyporesponder: Vadadustat 600 mg
Number analyzed (Participants) | 32 | 30 | 14 | 21 | 17 | 5
Hours
  Week 1 | 2.08 [0.00 to 11.50] | 2.72 [1.83 to 5.03] | 3.48 [1.92 to 10.50] | 3.50 [1.58 to 9.00] | 2.00 [1.75 to 5.03] | 3.28 [1.83 to 4.50]
  Week 1 +1 (Day 8): number analyzed (Participants) | 30 | 30 | 14 | 21 | 13 | 5
  Week 1 +1 (Day 8) | 3.28 [1.75 to 6.75] | 2.11 [0.00 to 5.23] | 3.33 [1.80 to 5.00] | 3.30 [0.00 to 5.00] | 2.17 [1.75 to 5.05] | 3.42 [1.80 to 4.50]
  Week 11: number analyzed (Participants) | 12 | 15 | 5 | 4 | 8 | 0
  Week 11 | 3.23 [0.00 to 4.50] | 3.50 [1.75 to 10.83] | 3.50 [2.00 to 4.67] | 2.03 [1.75 to 3.63] | 2.11 [1.80 to 5.00] |
  Week 13: number analyzed (Participants) | 0 | 4 | 1 | 0 | 2 | 0
  Week 13 |  | 1.98 [1.75 to 5.00] | 4.25 [4.25 to 4.25] |  | 2.04 [1.97 to 2.12] |

26. Secondary Outcome: Geometric Mean Elimination Rate Constant (λz) of Vadadustat Following a Single Dose
Description: Blood samples were collected from participants at defined time points for the assessment of λz of Vadadustat following a single dose.
Time Frame: as for outcome 22
Population: as for outcome 22
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1/hour
Arm/Group | Low Dose of Epoetin Alfa: Vadadustat 300 mg | Low Dose of Epoetin Alfa: Vadadustat 450 mg | High Dose of Epoetin Alfa: Vadadustat 300 mg | High Dose of Epoetin Alfa: Vadadustat 450 mg | High Dose of Epoetin Alfa: Vadadustat 600 mg | ESA Hyporesponder: Vadadustat 600 mg
Number analyzed (Participants) | 17 | 17 | 8 | 8 | 6 | 2
1/hour
  Week 1: number analyzed (Participants) | 17 | 17 | 7 | 8 | 5 | 2
  Week 1 | 0.0797 (38.7) | 0.0665 (50.5) | 0.0560 (41.6) | 0.0681 (32.7) | 0.0608 (46.9) | 0.0771 (8.9)
  Week 1 +1 (Day 8): number analyzed (Participants) | 13 | 16 | 8 | 8 | 6 | 2
  Week 1 +1 (Day 8) | 0.0720 (44.2) | 0.0615 (70.0) | 0.0714 (53.9) | 0.0469 (72.2) | 0.0469 (74.4) | 0.0594 (4.5)
  Week 11: number analyzed (Participants) | 6 | 6 | 2 | 1 | 3 | 0
  Week 11 | 0.0925 (65.5) | 0.0687 (26.5) | 0.124 (92.0) | 0.175 (NA) — Dispersion data are not available for a single participant | 0.116 (15.9) |
  Week 13: number analyzed (Participants) | 0 | 1 | 0 | 0 | 1 | 0
  Week 13 |  | 0.0632 (NA) — Dispersion data are not available for a single participant |  |  | 0.138 (NA) — Dispersion data are not available for a single participant |

27. Secondary Outcome: Geometric Mean Apparent Total Body Clearance (CLss/F) of Vadadustat Following a Single Dose
Description: Blood samples were collected from participants at defined time points for the assessment of CLss/F of Vadadustat following a single dose.
Time Frame: as for outcome 23
Population: as for outcome 22
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters per hour
Arm/Group | Low Dose of Epoetin Alfa: Vadadustat 300 mg | Low Dose of Epoetin Alfa: Vadadustat 450 mg | High Dose of Epoetin Alfa: Vadadustat 300 mg | High Dose of Epoetin Alfa: Vadadustat 450 mg | High Dose of Epoetin Alfa: Vadadustat 600 mg | ESA Hyporesponder: Vadadustat 600 mg
Number analyzed (Participants) | 29 | 28 | 13 | 21 | 13 | 5
liters per hour
  Week 1: number analyzed (Participants) | 27 | 23 | 11 | 19 | 12 | 5
  Week 1 | 0.888 (63.8) | 0.869 (71.1) | 0.877 (81.7) | 0.744 (54.5) | 0.763 (36.6) | 1.29 (80.9)
  Week 1 +1 (Day 8) | 1.04 (76.6) | 0.967 (80.8) | 0.968 (94.7) | 0.795 (41.1) | 0.708 (54.8) | 1.55 (112.4)
  Week 11: number analyzed (Participants) | 11 | 14 | 5 | 4 | 8 | 0
  Week 11 | 0.872 (53.5) | 1.33 (282.0) | 0.747 (70.8) | 1.00 (68.2) | 1.02 (52.5) |

28. Secondary Outcome: Geometric Mean Apparent Volume of Distribution (Vz/F) of Vadadustat Following a Single Dose
Description: Blood samples were collected from participants at defined time points for the assessment of Vz/F of Vadadustat following a single dose.
Time Frame: as for outcome 23
Population: as for outcome 22
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | Low Dose of Epoetin Alfa: Vadadustat 300 mg | Low Dose of Epoetin Alfa: Vadadustat 450 mg | High Dose of Epoetin Alfa: Vadadustat 300 mg | High Dose of Epoetin Alfa: Vadadustat 450 mg | High Dose of Epoetin Alfa: Vadadustat 600 mg | ESA Hyporesponder: Vadadustat 600 mg
Number analyzed (Participants) | 16 | 15 | 8 | 8 | 6 | 2
Liters
  Week 1: number analyzed (Participants) | 16 | 13 | 7 | 8 | 5 | 2
  Week 1 | 10.9 (36.2) | 14.3 (53.4) | 13.7 (69.7) | 12.1 (38.6) | 13.8 (16.7) | 15.8 (56.9)
  Week 1 +1 (Day 8): number analyzed (Participants) | 13 | 15 | 8 | 8 | 6 | 2
  Week 1 +1 (Day 8) | 12.5 (36.6) | 13.7 (41.0) | 17.4 (50.4) | 15.3 (67.4) | 15.6 (27.2) | 12.4 (35.8)
  Week 11: number analyzed (Participants) | 5 | 6 | 2 | 1 | 3 | 0
  Week 11 | 10.2 (28.7) | 10.7 (37.6) | 10.1 (10.3) | 8.24 (NA) — Dispersion data are not available for a single participant | 8.76 (18.9) |

ADVERSE EVENTS:
Time Frame: Up to Week 24 (from first dose of study drug to last dose + 4 weeks of follow-up)
Description: TEAEs, defined as AEs that began (or pre-existing AEs that worsened) on or after the first dose through each participant's last participation date, are reported. Safety Population: all participants in the Randomized Population who received at least 1 dose of study drug. Analysis of this population was based on actual treatment received. One participant randomized to the Low Dose of Epoetin Alfa: Vadadustat 300 mg arm inadvertently received 450 mg of Vadadustat.
Arm/Group | Low Dose of Epoetin Alfa: Vadadustat 300 mg | Low Dose of Epoetin Alfa: Vadadustat 450 mg | Low Dose of Epoetin Alfa: Epoetin Alfa | High Dose of Epoetin Alfa: Vadadustat 300 mg | High Dose of Epoetin Alfa: Vadadustat 450 mg | High Dose of Epoetin Alfa: Vadadustat 600 mg | High Dose of Epoetin Alfa: Epoetin Alfa | ESA Hyporesponder: Vadadustat 600 mg | ESA Hyporesponder: Epoetin Alfa
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/35 | 0/23 | 1/18 | 1/21 | 1/21 | 1/13 | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 9/34 | 7/35 | 5/23 | 8/18 | 6/21 | 10/21 | 5/13 | 4/5 | 3/5
Other Adverse Events (participants affected / at risk) | 11/34 | 20/35 | 10/23 | 9/18 | 9/21 | 10/21 | 8/13 | 4/5 | 2/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Dose of Epoetin Alfa: Vadadustat 300 mg (N=34) | Low Dose of Epoetin Alfa: Vadadustat 450 mg (N=35) | Low Dose of Epoetin Alfa: Epoetin Alfa (N=23) | High Dose of Epoetin Alfa: Vadadustat 300 mg (N=18) | High Dose of Epoetin Alfa: Vadadustat 450 mg (N=21) | High Dose of Epoetin Alfa: Vadadustat 600 mg (N=21) | High Dose of Epoetin Alfa: Epoetin Alfa (N=13) | ESA Hyporesponder: Vadadustat 600 mg (N=5) | ESA Hyporesponder: Epoetin Alfa (N=5)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nephrogenic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute left ventricular failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Incarcerated inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Incarcerated umbilical hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Catheter site thrombosis (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Liver injury (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gangrene (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Localised infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arteriovenous graft thrombosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Facial paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertensive encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metabolic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subcapsular renal haematoma (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nipple pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Uterine mass (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreas transplant (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Accelerated hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertensive crisis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertensive urgency (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Subclavian artery stenosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Dose of Epoetin Alfa: Vadadustat 300 mg (N=34) | Low Dose of Epoetin Alfa: Vadadustat 450 mg (N=35) | Low Dose of Epoetin Alfa: Epoetin Alfa (N=23) | High Dose of Epoetin Alfa: Vadadustat 300 mg (N=18) | High Dose of Epoetin Alfa: Vadadustat 450 mg (N=21) | High Dose of Epoetin Alfa: Vadadustat 600 mg (N=21) | High Dose of Epoetin Alfa: Epoetin Alfa (N=13) | ESA Hyporesponder: Vadadustat 600 mg (N=5) | ESA Hyporesponder: Epoetin Alfa (N=5)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Nephrogenic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bundle branch block right (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diastolic dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Left atrial enlargement (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Right atrial enlargement (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Systolic dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 3 (3) | 4 (5) | 4 (4) | 2 (3) | 4 (4) | 1 (1) | 1 (1) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ulcer haemorrhage (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acarodermatitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Localised infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nail infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 2 (2) | 2 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Graft thrombosis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transfusion reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vascular pseudoaneurysm ruptured (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypovolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Costovertebral angle tenderness (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Uterine haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Uraemic pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 0 (0)
Hypovolaemic shock (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Shock haemorrhagic (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vascular calcification (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Conclusions were drawn from results of the Main Study (n=165). As the sample size in the Erythropoiesis-stimulating Agent (ESA) Hyporesponder Parallel Study (n=10) was small in both the Vadadustat and Epoetin Alfa treatment groups, these results did not allow to meaningful interpretation of the data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-06-27): https://cdn.clinicaltrials.gov/large-docs/27/NCT03799627/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-02): https://cdn.clinicaltrials.gov/large-docs/27/NCT03799627/SAP_001.pdf